CLINICAL TRIAL: NCT02028416
Title: Protocol for Comparison of Two Different Regimens of Rabbit ATG-Fresenius With Cyclosporin in the Treatment of Acquired Aplastic Anaemia
Brief Title: Comparison of Two Different Doses of Rabbit ATG-Fresenius With Cyclosporin in the Treatment of Acquired Aplastic Anaemia
Acronym: ATG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Institute of Blood Disease Center, Pakistan (Other)
Responsible Party: Principal Investigator, MEHWESH TAJ, comparisor of two different regimens of AtG in Acquired Aplastic Anemia, National Institute of Blood Disease Center, Pakistan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIBD2571975
Record Dates: First submitted 2014-01-02; First posted 2014-01-07 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-04

CONDITIONS: Aplastic Anemia
Keywords: pancytopenia; aplastic anemia; ATG; Cyclosporin
MeSH Terms: conditions — Anemia, Aplastic; Pancytopenia | interventions — thymoglobulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ATG-Fresenius 3 Days (Active Comparator): In one group Injection ATG-Fresenius will be given @ 10mg/kg will be given for 3 days along with Capsule Cyclosporin 5mg/kg for 6 months followed by very slow tapering of dose
  Interventions: Drug: ATG-fresenius
- ATG-Fresenius 5 Days (Experimental): In other arm injection ATG will be given @10mg/Kg for 5 days (different dose regimen, according to the randomization) with capsule Cyclosporin@5mg/Kg (same dose) for 6 months followed by very slow tapering. There is a difference of days of treatment received i-e 5 days.
  Interventions: Drug: ATG-fresenius

INTERVENTIONS:
Drug: ATG-fresenius — we will create 2 arms as per randomization table. Both arms will receive ATG-Fresenius but with 2 different regimens.
  the first arm will receive ATG-F @10mg/kg for 3 days and second arm will receive ATG-F same dose but for 5 days
  Other Names: Rabbit ATG; ATG-F

SUMMARY:
Acquired Aplastic anemia is one of the most frequent reason of bone marrow failure in East (Pakistan).

* The first treatment option is Allogenic Bone Marrow transplantation which is an expansive treatment option and also require a full matched HLA identical donor, hence hardly 25% of our affected patients get opportunity for BMT.
* The second line treatment option caters a large chunk of patients (severe and non-severe AA) along with those who lack HLA identical donor.

Previously many protocols had been used in past for ATG+CsA Treatment, this treatment protocol especially addresses the two different regimens of ATG to study its efficacy, durability and long-term effects. Following doses would be used:

* CsA+ATG @ 10mg/kg for 3 days
* CsA+ATG @ 10mg/kg for 5 days

DETAILED DESCRIPTION:
Aplastic Anaemia (AA) is characterized by pancytopenia with hypo-cellular bone marrow in the absence of dysplasia, infiltration or fibrosis. The recommended first-line treatment options include Allogenic Bone Marrow Transplantation with HLA matched sibling donor. However, due to non-availability HLA matched identical sibling donor or due to other co-morbids and age, second choice of treatment is Anti Thymocyte Globulin (ATG) and Cyclosporin (CsA).

Rabbit ATG (Fresenius) has never been tested for the treatment of aplastic anaemia in Pakistani population before. We propose this investigator initiated trial which will will compare two different protocols of Rabbit ATG-Fresenius, 10mg/kg for 3 days and 10mg/kg for 5 days along with CsA in Pakistani patients suffering from AA. The subjects will be Non-severe (NSAA) and severe AA (SAA) who are not the eligible candidate for Allogenic Bone Marrow Transplantation. Patients will be randomized into two equal arms with same biological characteristics. Both arms will be treated with ATG-Fresenius and CsA in same doses with two different duration of treatment. They will later continue with CsA for at least 12 months and if response achieved, will be tapered more slowly over next 6 months.

The primary end point is to document the number of doses required by each of the two dose schedule to produce a response, achieve a nadir absolute lymphocyte count of 200 cmm. Secondary endpoints are short term safety of ATG-Fresenius, change in absolute neutrophil count from the baseline in both arms, change in platelet count from the baseline, change in absolute reticulocyte count, Number of blood units required till 8 weeks and 26 weeks, Number of platelet doses required till 8 weeks and 26 weeks, relapse, response rates at 6 and 12 months, clonal evolution to PNH, myelodysplasia or acute leukaemia. Long-course CsA will be assessed separately for its efficacy in reducing late events of relapse and evolution by comparison to historical control data.

ELIGIBILITY:
Inclusion Criteria:

i. Severe aplastic anemia characterized by: Bone marrow cellularity <30% (excluding lymphocytes) AND

At least two of the following:

a. Absolute neutrophil count < 500/ uL b. Platelet count < 20,000/ uL c. Absolute reticulocyte count <60,000/ uL i. Age > 2 years old ii. Weight > 9 kg

Exclusion Criteria:

i. Diagnosis of Fanconi's anemia ii. Evidence of a clonal disorder on cytogenetics. Patients with very severe neutropenia (ANC < 200 /uL) will be excluded iii. Failure of BMT iv. Prior immunosuppressive therapy with ATG, ALG, alemtuzumab, or high dose cyclophosphamide v. Infection not adequately responding to appropriate therapy vi. Serologic evidence of HIV infection vii. Failure to discontinue the herbal supplements or Other alternative approach of treatment within 2 weeks of enrolment viii. Moribund status or concurrent hepatic, renal, cardiac, neurologic, pulmonary, infectious, or metabolic disease of such severity that it would preclude the patient's ability to tolerate protocol therapy, or that death within 7-10 days is likely ix. History of carcinoma that is not considered cured (except local cervical, basal cell, or squamous cell) x. Current pregnancy, or unwillingness to take oral contraceptives or refrain from pregnancy if of childbearing potential xi. Not able to understand the investigational nature of the study or give informed consent

Ages: 2 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-09; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
absolute blood counts not meeting the criteria of Aplastic Anemia | 6 months
  Response is defined as blood counts no longer meeting the standard ("Camitta") criteria for severe pancytopenia in SAA, equivalent to 2 of the following values obtained on 2 serial blood count measurement at least one week apart at landmark time points (3, 6, and 12 months) .
  -To document the number of doses required by each of the two dose schedule to produce a rise in neutrophils and platelet count to achieve a nadir absolute lymphocyte count of 200 cmm Absolute neutrophil count > 500/ microL Platelet count > 20,000/ microL Reticulocyte count > 60,000/ microL

SECONDARY OUTCOMES:
transfusion dependency after ATG treatment | 2 years
  To document the short term safety of ATG-Fresenius at 8 weeks,12 weeks and then at 26 weeks in each arm
  * Number of blood units required till 8 weeks and 26 weeks
  * Number of platelet doses required till 8 weeks and 26 weeks
sustained improvement of blood counts post ATG | 2years
  To document the the change in absolute neutrophil, reticulocyte counts and platelet count from the baseline in each arm at 8 weeks, 12 weeks and then at 26 weeks
short-term safety of ATG and clonal evolution | 26 weeks
  to document the short term safety of ATG and development of any clonal evolution to PNH, myelodysplasia or acute leukaemia in patient
response rates of ATG treatment | 2 years
  to document the response rates of treatment with ATG+ Cyclosporin in patients with non-severe and severe Aplastic anemia at 6,12 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: TAHIR S SHAMSI, MBBS,FRCPath, Principal Investigator — NATIONAL INSTITUTE OF BLOOD DISEASES AND BONE MARROW TRANSPLANTATION; MEHWESH TAJ, MBBS, FCPS, Study Director — NATIONAL INSTITUTE OF BLOOD DISEASES AND BONE MARROW TRANSPLANTATION; UZMA RIZVI, MBBS, Study Chair — NATIONAL INSTITUTE OF BLOOD DISEASES AND BONE MARROW TRANSPLANTATION
Locations (1):
- National Institute of Blood Diseases and Bone Marrow Transplantation, Karachi, Pakistan, Pakistan

IPD SHARING:
Plan to Share IPD: No
All data saved at research department of NIBD under supervision of PI